CLINICAL TRIAL: NCT06810115
Title: Incidence and Clinical Significance of Respiratory Viral Infections in Patients with Multiple Myeloma
Brief Title: Respiatory Viral Infections in Patients with Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Polona Novak, Polona Novak, MD, University Medical Centre Ljubljana
Other Study IDs: 83/03/15
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2015-03

CONDITIONS: Multiple Mieloma; Respiratory Viral Infections
Keywords: Respiratory viral infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Viral PCR testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient with multiple myeloma
  Interventions: Other: Viral PCR test

INTERVENTIONS:
Other: Viral PCR test — Viral PCR test regardles of symptoms

SUMMARY:
Respiratory viruses are known to be a major cause of morbodity in multiple myeloma patients but prospective long-term sudies are lacking. We analysed 219 multiple myeloma patients that had 554 nasopharingeal swabs with 58 documented viral episodes. Respiratory viruses studied were rhinovirus, enterovirus, parainflienza, respirator, syncytial virus, metapneumovirus, coronavirus, bocavirus, influenza A, influenza B. Clinical data were extracted from a prospectively entered database, medical records were reviewed. We have prospectively studiend patients until May 2019 when we gathered survival data. Lastly because of Covid-19 pandemic when almost no other viral infections were isolated, we analysed clinical course of respiratory infections in patients with multiple myeloma after the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma

Exclusion Criteria:Other hematological malignancies

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with multiple myeloma on observation/receiving treatment at outpatient clinuc
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Number of respiratory viral infections in patirnts with multiple myeloma | 1 year

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blimark C, Holmberg E, Mellqvist UH, Landgren O, Bjorkholm M, Hultcrantz M, Kjellander C, Turesson I, Kristinsson SY. Multiple myeloma and infections: a population-based study on 9253 multiple myeloma patients. Haematologica. 2015 Jan;100(1):107-13. doi: 10.3324/haematol.2014.107714. Epub 2014 Oct 24. PMID 25344526